CLINICAL TRIAL: NCT00884598
Title: Cilengitide (EMD121974) in Combination With Whole Brain Radiotherapy in Patients With Brain Metastases From Lung Cancer - a Single-center, Open-label Phase I Study
Brief Title: Cilengitide and Whole-Brain Radiation Therapy in Treating Patients With Brain Metastases From Lung Cancer
Acronym: CIRAB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Principal Investigator, Frederik Wenz, Prof. Christian Manegold, Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000636508; HUMCM-CIRAB; EUDRACT-2008-004573-17
Record Dates: First submitted 2009-04-18; First posted 2009-04-21 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Brain and Central Nervous System Tumors; Lung Cancer
Keywords: adult tumors metastatic to brain; extensive stage small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Central Nervous System Neoplasms; Lung Neoplasms; Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cilengitide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cilengitide (Experimental)
  Interventions: Drug: cilengitide; Other: pharmacological study; Radiation: radiation therapy

INTERVENTIONS:
Drug: cilengitide
Other: pharmacological study
Radiation: radiation therapy

SUMMARY:
RATIONALE: Cilengitide may stop the growth of brain metastases by blocking blood flow to the tumor. Radiation therapy uses high energy X-rays to kill tumor cells. Giving cilengitide together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of cilengitide when given together with whole-brain radiation therapy in treating patients with brain metastases from lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Primary

  * To assess the safety and tolerability of daily cilengitide by determining its dose-limiting toxicity and maximum-tolerated dose when combined with concomitant fractionated whole-brain radiation therapy in patients with brain metastases from lung cancer.
* Secondary

  * To collect evidence of the best overall response rate, overall survival, brain-specific progression-free survival, and tumor-specific progression-free survival of these patients.
  * To collect evidence of changes in functional MRI imaging studies at 6 and 12 weeks after initiation of therapy.
  * To collect evidence of early response by functional MRI (ASL technique) on days 1, 4, and 12, immediately before and after the administration of cilengitide.
  * To collect evidence of changes in neurological and neurocognitive function tests at 6 and 12 weeks after initiation of therapy.
  * To further evaluate the safety and toxicity of the combination of cilengitide and whole-brain radiation therapy.
  * To further evaluate the pharmacokinetics of cilengitide administered daily.

OUTLINE:

Patients receive oral cilengitide once daily and undergo whole-brain radiotherapy on the same days. Treatment continues for 2 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection on days 1, 4, 5, and 12 for pharmacokinetic studies.

After completion of study treatment, patients are followed for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed lung cancer (small cell or non-small cell lung cancer)
* Patient must be eligible for whole-brain radiotherapy
* Presence of brain metastasis (single or multiple, synchronous or metachronous) from lung cancer not amenable to surgery or radiosurgery (presence of metastases at any other site is allowed)
* No leptomeningeal metastasis or known subarachnoid spread of tumor

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 (ECOG PS 2 allowed if due to the presence of cerebral metastases and not due to a high peripheral-tumor load or other reasons)
* Life expectancy ≥ 3 months
* Adequate hematologic function
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* AST, ALT, and alkaline phosphatase < 2.5 times ULN
* Creatinine clearance > 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No history of acute or chronic renal disease
* No other malignancies treated within the past 5 years, except adequately treated carcinoma in situ of the cervix or basal cell carcinoma of the skin
* No uncontrolled hypertension
* No history of coagulation disorder associated with bleeding or recurrent thrombotic events
* No peptic ulcer disease within the past 6 months
* No congestive heart failure, high risk for uncontrolled arrhythmia, or history of clinically significant coronary heart disease
* No known alcohol or drug abuse
* No other significant or acute concomitant disease
* No dementia or altered mental status

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent corticosteroids allowed if the dosing regimen has ben stable ≥ 5 days
* Concurrent anticonvulsants allowed if the dosing regimen has been stable for the past week
* More than 30 days since prior participation in another clinical trial
* No concurrent anticoagulation with vitamin K antagonists, therapeutic-dose anticoagulation with heparin resulting in prolonged PTT, or therapeutic-dose anticoagulation with low molecular weight heparin (low-dose [i.e. prophylactic], low molecular weight heparins allowed)
* No prior whole-brain radiation or radiosurgery
* No prior antiangiogenic therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 12 days
  (i) Any grade III-IV non-hematological toxicity as defined by CTCAE, version 3.0, with the exclusion ofalopecia, nausea, vomiting, and fever that can be rapidly contolled with appropriate measures; (ii) absolute neutrophil count (ANC)<0.5x10'/L lasting for >7days; (iii) febrile neutropenia defined as ANC <1.0x10'/L and fever >38.5°C; (iv) platelets <25x10'/L or thrombocytopenic bleeding requiring transfusion; and (v) severe hypotension requiring dopamine administration.
Maximum-tolerated dose | 12 days
  5 planned steps to be tested: 100, 250, 500, 750, to 1000mg; the highest dose at which one or no DLT will have been observed among 6 patients

SECONDARY OUTCOMES:
Overall response rate | 12 weeks
  Any response to treatment
Overall survival | 1 year
  Death as event, Kaplan-Meier (KM)
Brain-specific progression-free survival (PFS) | 1 year
  Every recurrence within the brain or death is an event, Kaplan-Meier (KM)
Tumor-specific PFS | 1 year
  Every tumor related event or death will be counted, Kaplan-Meier (KM)
Changes in functional MRI imaging (time to peak) at 6 and 12 weeks | 12 weeks
  time-to-peak measurements
Changes in functional MRI imaging (blood flow) at 6 and 12 weeks | 12 weeks
  blood flow measurements
Changes in functional MRI imaging (blood volume changes) at 6 and 12 weeks | 12 weeks
  blood volume changes during functional MRI
Evidence of early response by functional MRI on days 1, 4, and 12 | 12 days
  (ASL technique) on day 1,4 and 12, immediately before and after the administration of cilengitide.
Changes of neurocognitive function tests (intelligence) at 6 and 12 weeks | 12 weeks
  Intelligence was measured with a multiple-choice test of vocabulary knowledge.
Changes of neurocognitive function tests (memory figures) at 6 and 12 weeks | 12 weeks
  Memory was tested by aims of "Medical College of Georgia Complex Figures"
Changes of neurocognitive function tests (memory verbal) at 6 and 12 weeks | 12 weeks
  Memory was tested by aims of "Rea Auditory Verbal Learning Test - German Version"
Changes of neurocognitive function tests (perception) at 6 and 12 weeks | 12 weeks
  Perception was assessed by the "Digit Symbol Substitution Test"
Changes of neurocognitive function tests (attention/alertness) at 6 and 12 weeks | 12 weeks
  Attention was tested by "Alertness"
Changes of neurocognitive function tests (attention) at 6 and 12 weeks | 12 weeks
  Attention was tested by "Divided Attention"
Changes of neurocognitive function tests (attention speaking) at 6 and 12 weeks | 12 weeks
  Attention was tested by "Go,A.lo-Go".
Fatigue at 6 and 12 weeks | 12 weeks
  "Functional Assessment of Cancer Therapy - Fatigue Subscale" measured in points (range 0-52)
Anxiety/depression at 6 and 12 weeks | 12 weeks
  "Hospital Anxiety and Depression Scale - German Version"
Activities of daily living (Barthel) at 6 and 12 weeks | 12 weeks
  "Barthel Activities of Daily Living Index" measured in points (range 0-100)
Activities of daily living (instrumental) at 6 and 12 weeks | 12 weeks
  "lnstrumental Activities of Daily Living Scale" measured in points (range 0-8)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Manegold, MD, Principal Investigator — University Medical Center Mannheim
Locations (1):
- University Medical Center, Department of Surgery, Mannheim, Germany